CLINICAL TRIAL: NCT07206056
Title: TulmiSTAR-01: A Two-part, Phase I Dose Escalation and Expansion Followed by a Randomized, Open-label Multicenter, Phase II Study to Assess the Safety and Efficacy of the Combination of Tulmimetostat (DZR123) and JSB462 (Luxdegalutamide) vs Standard of Care in Patients With Progressive Metastatic Castrate Resistant Prostate Cancer
Brief Title: An Open-label Dose Escalation and Expansion, Followed by a Phase II Study of Tulmimetostat (DZR123) and JSB462 (Luxdegalutamide) in Patients With Progressive Metastatic Castrate Resistant Prostate Cancer (mCRPC) (TulmiSTAR-01)
Acronym: TulmiSTAR-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDZR123A12107; 2025-521880-10-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-09-17; First posted 2025-10-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Progressive Metastatic Castrate Resistant Prostate Cancer
Keywords: metastatic castrate resistant prostate cancer (mCRPC); tulmimetostat (DZR123); luxdegalutamide (JSB462); Androgen Deprivation Therapy (ADT); Standard of care (SoC); TulmiSTAR-01
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Part 1a (dose escalation): Participants will be assigned to cohorts to receive study treatment (tulmimetostat and JSB462) at different provisional dose levels.
  Part 1b (dose expansion and optimization): Participants will be randomized in a ratio and receive study treatment as:
  * Arm A: Tulmimetostat Dose 1 QD + JSB462 QD
  * Arm B: Tulmimetostat Dose 2 QD + JSB462 QD
  Part 2: Participants will be randomized in a ratio and receive study treatment as:
  * Arm 1: Tulmimetostat RP2D QD + JSB462 (either Dose 1 or Dose 2 QD)
  * Arm 2 (Control): SoC (ARPI, chemotherapy, Pluvicto) at the discretion of the investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part 1a: Cohort DL1A (Experimental): Tulmimetostat DL1 QD + JSB462 Dose 1 QD
  Interventions: Drug: Tulmimetostat DL1 QD; Drug: JSB462 Dose 1 QD
- Part 1a: Cohort DL1B (Experimental): Tulmimetostat DL1 QD + JSB462 Dose 2 QD
  Interventions: Drug: Tulmimetostat DL1 QD; Drug: JSB462 Dose 2 QD
- Part 1a: Cohort DL2A (Experimental): Tulmimetostat DL2 QD + JSB462 Dose 1 QD
  Interventions: Drug: Tulmimetostat DL2 QD; Drug: JSB462 Dose 1 QD
- Part 1a: Cohort DL2B (Experimental): Tulmimetostat DL2 QD + JSB462 Dose 2 QD
  Interventions: Drug: Tulmimetostat DL2 QD; Drug: JSB462 Dose 2 QD
- Part 1a: Cohort DL3A (Experimental): Tulmimetostat DL3 QD + JSB462 Dose 1 QD
  Interventions: Drug: Tulmimetostat DL3 QD; Drug: JSB462 Dose 1 QD
- Part 1a: Cohort DL3B (Experimental): Tulmimetostat DL3 QD + JSB462 Dose 2 QD
  Interventions: Drug: Tulmimetostat DL3 QD; Drug: JSB462 Dose 2 QD
- Part 1b : Arm A (Experimental): Tulmimetostat Dose 1 QD + JSB462 QD
  Interventions: Drug: Tulmimetostat Doses 1 or 2 QD; Drug: JSB462 QD
- Part 1b: Arm B (Experimental): Tulmimetostat Dose 2 QD + JSB462 QD
  Interventions: Drug: Tulmimetostat Doses 1 or 2 QD; Drug: JSB462 QD
- Part 2: Arm 1 (Experimental): Tulmimetostat RP2D QD + JSB462 QD
  Interventions: Drug: Tulmimetostat RP2D QD; Drug: JSB462 QD
- Part 2: Arm 2 (Active Comparator): Standard of Care at the discretion of the investigator
  Interventions: Drug: Standard of Care (SoC)

INTERVENTIONS:
Drug: Tulmimetostat DL1 QD — Part 1a (dose escalation):
  Doses of tulmimetostat beyond DL1 once a day (QD) will be opened depending on outcome of Dose Escalation Meetings (DEM(s))
  Other Names: DZR123
  Arms: Part 1a: Cohort DL1A; Part 1a: Cohort DL1B
Drug: Tulmimetostat DL2 QD — Part 1a (dose escalation):
  Doses of tulmimetostat beyond DL1 once a day (QD) will be opened depending on outcome of Dose Escalation Meetings (DEM(s))
  Other Names: DZR123
  Arms: Part 1a: Cohort DL2A; Part 1a: Cohort DL2B
Drug: Tulmimetostat DL3 QD — Part 1a (dose escalation):
  Doses of tulmimetostat beyond DL1 once a day (QD) will be opened depending on outcome of Dose Escalation Meetings (DEM(s))
  Other Names: DZR123
  Arms: Part 1a: Cohort DL3A; Part 1a: Cohort DL3B
Drug: Tulmimetostat Doses 1 or 2 QD — Part 1b (dose expansion and optimization):
  tulmimetostat doses 1 or 2 QD
  Other Names: DZR123
  Arms: Part 1b : Arm A; Part 1b: Arm B
Drug: Tulmimetostat RP2D QD — Part 2:
  tulmimetostat Recommended Phase 2 Dose (RP2D) QD
  Other Names: DZR123
  Arms: Part 2: Arm 1
Drug: JSB462 Dose 1 QD — JSB462 Dose 1 QD
  Other Names: luxdegalutamide
  Arms: Part 1a: Cohort DL1A; Part 1a: Cohort DL2A; Part 1a: Cohort DL3A
Drug: JSB462 Dose 2 QD — JSB462 Dose 2 QD
  Other Names: luxdegalutamide
  Arms: Part 1a: Cohort DL1B; Part 1a: Cohort DL2B; Part 1a: Cohort DL3B
Drug: JSB462 QD — The dose of JSB462 QD will be determined based on the totality of data from Part 1a
  Other Names: luxdegalutamide
  Arms: Part 1b : Arm A; Part 1b: Arm B; Part 2: Arm 1
Drug: Standard of Care (SoC) — Androgen Receptor Pathway Inhibitors (ARPI), chemotherapy or Pluvicto (AAA617) at the discretion of the investigator
  Arms: Part 2: Arm 2

SUMMARY:
This is a two-part, Phase I/II, open-label, global, multicenter study assessing the safety and efficacy of the combination of tulmimetostat (DZR123) and JSB462 (luxdegalutamide) versus standard of care in participants with progressive metastatic castrate resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
The Phase 1 study, comprised of Parts 1a and 1b, aims to assess the safety and tolerability of the combination of tulmimetostat and JSB462:

1. Part 1a is the parallel dose escalation that aims to determine the recommended dose(s) of tulmimetostat and JSB462, in combination, for further exploration.
2. Part 1b is the dose expansion/optimization that aims to determine the recommended dose of the combination for Phase II.

The purpose of the Phase II study (Part 2) is to compare the combination of tulmimetostat with JSB462 in terms of the biochemical response as assessed by PSA50 compared to the standard of care (SoC) in adult men with progressive, taxane-naive mCRPC.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is an adult man ≥ 18 years of age.
* Participant must have histologically and/or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine or small cell features (current or prior biopsy of the prostate and/or metastatic site).
* Participant must have ≥ 1 metastatic lesion that is present on screening/baseline CT, MRI, or bone scan imaging obtained ≤ 28 days prior to start of treatment (Part 1a dose escalation) or randomization (Part 1b dose expansion and Part 2).
* Participant must have progressive mCRPC.
* Participant must have a castrate level of serum/plasma testosterone (< 50 ng/dL or < 1.7 nmol/L).
* Prior ARPI therapy:

  * Part 1a and 1b only: must have progressed on at least one prior second generation ARPI (abiraterone, enzalutamide, darolutamide, or apalutamide).
  * Part 2 only: must have progressed on one prior second generation ARPI (abiraterone, enzalutamide, darolutamide, or apalutamide).
* Prior chemotherapy:

  * Part 1a dose escalation only: may have received ≤ 2 prior lines of chemotherapy in CRPC setting. Note: Prior chemotherapy is permitted in the HSPC setting.
  * Part 1b dose expansion/optimization only: may have received up to one prior line of chemotherapy in CRPC setting. Note: Prior chemotherapy is permitted in the HSPC setting.
  * Part 2 only: Participants must be taxane-naïve in mCRPC setting; prior chemotherapy permitted in HSPC setting only

Key Exclusion Criteria:

* Previous treatment with any PRC2 inhibitor, including but not limited to EZH2 inhibitors, EZH2/1 inhibitors, or embryonic ectoderm development (EED) inhibitors.
* Previous treatment with a protein degrader compound that targets the AR.
* Known hypersensitivity or contraindication to any of the study treatment components or its excipients or to drugs of similar chemical classes.
* Treatment with any investigational agent within 28 days (or 5 half-lives, whichever is longer) prior to study entry.
* Previous treatment with radioligand therapy in the mCRPC setting, except in Part 1a where participants may have received RLT in mCRPC setting.
* Participants with evidence of mCRPC or biochemical recurrence / PSA only disease or asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy and with normal PSA for ≥ 1 year prior to study entry.
* Participants with a history of CNS metastases must have received therapy (surgery, radiotherapy, gamma knife) and be neurologically stable, asymptomatic, and not receiving corticosteroids for the purpose of maintaining neurologic integrity. Those with leptomeningeal disease are eligible if those areas have been treated, are stable, and no neurological impairment is present. For those with parenchymal CNS metastasis (or a history of CNS metastasis), baseline and subsequent radiological imaging must include evaluation of the brain with MRI (preferred) or CT with contrast.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult men with metastatic castrate resistant prostate cancer (mCRPC)
Enrollment: 188 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2029-10-29 (Estimated); Study Completion 2030-12-17 (Estimated)

PRIMARY OUTCOMES:
Part 1a: Dose-limiting toxicities (DLTs) | Up to 28 days
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness/injury, or concomitant medications that occurs within the first 28 days of treatment with tulmimetostat and JSB462 and meets any of the criteria specified in the protocol. The National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) version 5.0 will be used for all grading. For the purpose of dose-escalation decisions, DLTs will be considered and included in the Bayesian Logistic Regression Model (BLRM).
Part 1a and Part 1b: Incidence rate of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From date of randomization till 30 days safety fup, assessed up to approximately 14 months
  The analysis of adverse events will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Part 1a and Part 1b: Number of Participants with dose adjustments | From date of randomization till 30 days safety fup, assessed up to approximately 14 months
  The number of participants with dose adjustments (reductions, interruption, or permanent discontinuation) will be summarized by treatment arm.
Part 1a and Part 1b: Dose Intensity | From date of randomization till 30 days safety fup, assessed up to approximately 14 months
  Dose intensity (computed as the ratio of actual cumulative dose received and actual duration of exposure) and the relative dose intensity (computed as the ratio of dose intensity and planned dose intensity) will be summarized by means of descriptive statistics
Part 1a and Part 1b: Duration of exposure to each study drug | From date of randomization till 30 days safety fup, assessed up to approximately 14 months
  The duration of exposure (in months) to Tulmimetostat and JSB462 (Part 1a and Part 1b) will be summarized by means of descriptive statistics
Part 1b and Part 2: prostate-specific antigen 50 (PSA50) at Month 6 | Month 6
  PSA50 is defined as a PSA reduction of at least 50% from baseline at 6 months confirmed by a second PSA measurement ≥ 3 weeks later.

SECONDARY OUTCOMES:
Part 1a and Part 1b: Plasma concentrations of tulmimetostat and JSB462 | Cycle 1-2: Day 1 (predose/0 hour, 1 hour, 2 hours, 4 hours, 6 hours and 8 hours; Tulmimetostat only: 30 minutes and 3 hours). Cycle 1: Day 2 (24 hours), Days 8 and 15 (predose/0 hour and 2 hours). Cycles 3-5: Day 1 (predose/0 hour). 1 cycle = 28 days.
  Tulmimetostat and JSB462 pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels by treatment arms
Part 2: Plasma concentrations of tulmimetostat and JSB462 | Cycle 1 and 2: Day 1 (predose/0 hour and 2 hours). Cycles 3-5: Day 1 (predose/0 hour). 1 cycle = 28 days.
  Tulmimetostat and JSB462 pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels by treatment arms
Part 1a and Part 1b: AUC of tulmimetostat and JSB462 | Cycle 1-2: Day 1 (predose/0 hour, 1 hour, 2 hours, 4 hours, 6 hours and 8 hours; Tulmimetostat only: 30 minutes and 3 hours). Cycle 1: Day 2 (24 hours), Days 8 and 15 (predose/0 hour and 2 hours). Cycles 3-5: Day 1 (predose/0 hour). 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) and Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) will be listed and summarized using descriptive statistics.
Part 2: AUC of tulmimetostat and JSB462 | Cycle 1 and 2: Day 1 (predose/0 hour and 2 hours). Cycles 3-5: Day 1 (predose/0 hour). 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) and Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) will be listed and summarized using descriptive statistics.
Part 1a and Part 1b: Cmax of tulmimetostat and JSB462 | Cycle 1-2: Day 1 (predose/0 hour, 1 hour, 2 hours, 4 hours, 6 hours and 8 hours; Tulmimetostat only: 30 minutes and 3 hours). Cycle 1: Day 2 (24 hours), Days 8 and 15 (predose/0 hour and 2 hours). Cycles 3-5: Day 1 (predose/0 hour). 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Part 2: Cmax of tulmimetostat and JSB462 | Cycle 1 and 2: Day 1 (predose/0 hour and 2 hours). Cycles 3-5: Day 1 (predose/0 hour). 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Part 1b and Part 2: prostate-specific antigen 50 (PSA50) at 3, 9, and 12 months | Month 3, Month 9, Month 12
  PSA50 is defined as a PSA reduction of at least 50% from baseline at 3, 9, and 12 months confirmed by a second PSA measurement ≥ 3 weeks later.
Part 1b and Part 2: radiographic progression free survival (rPFS) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 15 months
  rPFS is defined as time between randomization and the first occurrence of disease progression as per PCWG3-modified RECIST v1.1 or death due to any cause
Part 1b and Part 2: overall survival (OS) | From date of randomization until date of death from any cause, assessed up to approximately 15 months
  OS is defined as the time between randomization to date of death due to any cause
Part 1b and Part 2: objective response (OR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 15 months
  OR is defined as a confirmed complete response (CR) or partial response (PR) per PCWG3-modified RECIST 1.1 as assessed by the investigator
Part 1b and Part 2: best overall response (BOR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 15 months
  BOR is defined as the best response per Prostate Cancer Working Group 3 (PCWG3)-modified RECIST 1.1 as assessed by the Investigator
Part 1b and Part 2: duration of response (DOR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 15 months
  DOR is defined as time between first documented CR/PR and disease progression or death due to any cause per PCWG3-modified RECIST 1.1 as assessed by the investigator
Part 1b and Part 2: time to first symptomatic skeletal event (TTSSE) | From randomization until the first occurrence of a new symptomatic bone fracture, spinal cord compression, tumor-related orthopedic surgery, radiation therapy for bone pain, or death, assessed up to 15 months.
  TTSSE is defined as time from randomization to the first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain or death from any cause, whichever occurs first.
Part 2: Incidence rate of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From date of randomization till 30 days safety fup, assessed up to approximately 15 months
  The analysis of adverse events will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Part 2: Number of Participants with dose adjustments | From date of randomization till 30 days safety fup, assessed up to approximately 15 months
  The number of participants with dose adjustments (reductions, interruption, or permanent discontinuation) will be summarized by treatment arm.
Part 2: Dose Intensity | From date of randomization till 30 days safety fup, assessed up to approximately 15 months
  Dose intensity (computed as the ratio of actual cumulative dose received and actual duration of exposure) and the relative dose intensity (computed as the ratio of dose intensity and planned dose intensity) will be summarized by means of descriptive statistics
Part 2: Duration of exposure to each study drug | From date of randomization till 30 days safety fup, assessed up to approximately 15 months
  The duration of exposure (in months) to Tulmimetostat and JSB462 / Standard of Care (SoC) of investigator's choice (Part 2) will be summarized within each strata by means of descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (4):
  - Sarah Cannon Research Institute, Denver, Colorado
  - Sarah Cannon Research Institute, Jacksonville, Florida
  - Wichita Urology Group PA, Wichita, Kansas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (2):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Liverpool
- Novartis Investigative Site, Vejle, Denmark
- Novartis Investigative Site, Bordeaux, France
- Novartis Investigative Site, Kuching, Sarawak, Malaysia
- Novartis Investigative Site, Poznan, Poland
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com